CLINICAL TRIAL: NCT01030406
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study to Assess the Relative Abuse Potential of Acurox Tablets in Non-Dependent Recreational Opioid Users
Brief Title: Study of the Relative Abuse Potential of Acurox Tablets in Non-Dependent Recreational Opioid Users
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acura Pharmaceuticals Inc. (Industry)
Collaborators: King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AP-ADF-114
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2010-03

CONDITIONS: Opioid Abuse
Keywords: Abuse Liability; Abuse Prevention; Abuse Resistance; Abuse Deterrence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Matching white tablets
Oversight: Data Monitoring Committee: No

ARMS (5):
- 40/0mg taken first (Active Comparator): 8x oxycodone/niacin 5/0mg tablets
  Interventions: Drug: 40/0mg taken first
- 80/0mg taken first (Active Comparator): 8x oxycodone/niacin 10/0mg tablets
  Interventions: Drug: 80/0mg taken first
- 40/240mg taken first (Experimental): 8x oxycodone/niacin 5/30mg tablets
  Interventions: Drug: 40/240mg taken first
- 80/480mg taken first (Experimental): 8x oxycodone/niacin 10/60mg tablets
  Interventions: Drug: 80/480mg taken first
- 0/0mg taken first (Placebo Comparator): Placebo
  Interventions: Drug: 0/0mg taken first

INTERVENTIONS:
Drug: 40/0mg taken first — 8x Oxycodone/Niacin 5/0mg tablets All arms taken with a 48 hour washout between doses
  Arms: 40/0mg taken first
Drug: 80/0mg taken first — 8x Oxycodone/Niacin 10/0mg tablets All arms taken with a 48 hour washout between doses
  Arms: 80/0mg taken first
Drug: 40/240mg taken first — 8x Oxycodone/Niacin 5/30mg tablets All arms taken with a 48 hour washout between doses
  Arms: 40/240mg taken first
Drug: 80/480mg taken first — 8x Oxycodone/Niacin 10/60mg tablets All arms taken with a 48 hour washout between doses
  Arms: 80/480mg taken first
Drug: 0/0mg taken first — Placebo All arms taken with a 48 hour washout between doses
  Arms: 0/0mg taken first

SUMMARY:
The primary objective of this study is to compare the relative abuse potential of two different doses of orally administered Acurox Tablets to orally administered immediate-release (IR) oxycodone HCl tablets in non-dependent recreational opioid users.

DETAILED DESCRIPTION:
In the tretament phase, 5 treatments administered were oxycodone HCl/niacin tablets as follows: (A) 40/0 mg, (B) 80/0 mg, (C) (40/240 mg, (D) 80/480 mg and (E) 0/0 mg. Each treatment was administered as a single dose of 8 tablets once a day at approximately the same time each day. All doses were given with water, and all 8 tablets were to be swallowed in 5 minutes. Doses were separated by 48 (± 1) hours. All subjects received each treatment in a randomized sequence using a Williams design.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female between 18 and 55 years old.
* Subject is in generally good health, including no history of pulmonary disease, and has a body mass index (BMI) within 18-33 kg/m2.
* Subject is a recreational opioid user (i.e., at least 10 occasions within the past 12 months, and at least 1 within the past 12 weeks) who is NOT physically dependent on opioids (per Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision [DSM-IV-TR]); is able to speak, read, and understand English; and will provide written informed consent.
* Subject has a minimum of a 6th grade reading level as determined by the Investigator or by the Rapid Estimation of Adult Literacy in Medicine (REALM).

Exclusion Criteria:

* History or current diagnosis of substance dependence (except nicotine and caffeine) and/or alcohol abuse according to the criteria of DSM-IV-TR.
* History or current diagnosis of neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, hematologic, pulmonary, or metabolic disease.
* Known allergy or history of hypersensitivity to oxycodone HCl, other opioids, or any component of Acurox Tablets.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Webster, MD, Principal Investigator — Lifetree Clinical Research
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 40/0mg Taken First: Ocycodone/Naicin 40/0mg Tablets
- 80/0mg Taken First: Oxycodone/Niacin 80/0mg tablets
- 40/240mg Taken First: Oxycodone?Niacin 40/240mg tablets
- 80/480mg Taken First: Oxycodone/Naicin 80/480mg
- 0/0mg Taken First: Placebo: Tablets
Period: Overall Study
Arm/Group | 40/0mg Taken First | 80/0mg Taken First | 40/240mg Taken First | 80/480mg Taken First | 0/0mg Taken First
Started | 10 | 10 | 10 | 10 | 9
Completed | 10 | 10 | 9 | 9 | 9
Not Completed | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Crossover design. Subjects took all drugs in randomized order with a 48 hour washout between doses
Groups:
- 40/0mg Taken First: oxycodone.naicin 40/0mg tablets
- 80/0mg Taken First: oxycodone.naicin 80/0mg tablets
- 40/240mg Taken First: oxycodone.naicin 40/240mg tablets
- 80/480mg Taken First: oxycodone.naicin 80/480mg tablets
- 0/0mg Taken First: Placebo Tablets
- Total: Total of all reporting groups
Arm/Group | 40/0mg Taken First | 80/0mg Taken First | 40/240mg Taken First | 80/480mg Taken First | 0/0mg Taken First | Total
Number analyzed (Participants) | 10 | 10 | 9 | 9 | 9 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 9 | 9 | 9 | 47
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 drop out; 1 protocol violation
  years | 23.9 (4.83) | 23.9 (4.83) | 23.9 (4.83) | 23.9 (4.83) | 23.9 (4.83) | 23.9 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 2 | 2 | 12
  Male | 7 | 7 | 7 | 7 | 7 | 35
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 9 | 9 | 47

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking at .5 Hours
Description: Drug Liking/Disliking Assessment on a 101 point bipolar visual analog scale (VAS) used to assess response to the question "Do you dislike or like the drug effect you are feeling now?" and anchored in the center with "Neither like nor dislike" (score of 50), on the left with "Dislike an awful lot" (score of 0) and on the right with "Like an awful lot" (score of 100).
Time Frame: Measure collected at 0.5 hours post-dose
Population: Per protocol completers
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 40/0mg: 8x Oxycodone/Naicin 5/0mg tablets
- 80/0mg: 8x Oxycodone/Naicin 10/0mg tablets
- 40/240mg: 8x Oxycodone/Naicin 5/30mg tablets
- 80/480mg: 8x Oxycodone/Naicin 10/60mg tablets
- 0/0mg: Placebo: Tablets
Arm/Group | 40/0mg | 80/0mg | 40/240mg | 80/480mg | 0/0mg
Number analyzed (Participants) | 46 | 46 | 46 | 46 | 46
score on a scale | 66.0 (16.44) | 74.7 (16.86) | 47.7 (19.96) | 40.9 (22.93) | 50.3 (2.28)

ADVERSE EVENTS:
Groups:
- 40/0mg; 80/0mg: Oxycodone hcl 40mg
- 40/240mg: Oxycodone hcl 40mg/niacin 240mg
- 80/480ng: Oxycodone hcl 80mg/niacin 480mg
Arm/Group | 40/0mg | 80/0mg | 40/240mg | 80/480ng | 0/0mg
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 37/49 | 46/49 | 47/49 | 49/49 | 3/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40/0mg (N=49) | 80/0mg (N=49) | 40/240mg (N=49) | 80/480ng (N=49) | 0/0mg (N=49)
Flushing (Vascular disorders) | 0 (0) | 3 (3) | 43 (43) | 46 (46) | 0 (0) — Flushing
Pruritis (Skin and subcutaneous tissue disorders) | 29 (29) | 34 (34) | 36 (36) | 39 (39) | 2 (2)
Somnolence (Nervous system disorders) | 17 (17) | 18 (18) | 13 (13) | 22 (22) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 6 (6) | 3 (3) | 6 (6) | 0 (0)
nausea (Gastrointestinal disorders) | 4 (4) | 18 (18) | 5 (5) | 17 (17) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 11 (11) | 4 (4) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No